CLINICAL TRIAL: NCT01031862
Title: A Pilot Study to Evaluate the Use of 3H Particulate Cholesterol as a Method to Study Reverse Cholesterol Transport in Humans
Brief Title: BMS Reverse Cholesterol Transport (RCT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 810035; CV 197-003
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: healthy volunteer; reverse cholesterol transport; RCT; 3H

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Other): 12 healthy volunteers
  Interventions: Other: 3H-Cholesterol

INTERVENTIONS:
Other: 3H-Cholesterol — A single dose of 25-50 μCi 3H free cholesterol -albumin complexes (containing approximately 0.1 - 0.3 mg of cholesterol) will be administered intravenously as a slow bolus injection within 1-2 minutes.

SUMMARY:
The purpose of this study is to investigate the use of radiolabeled particulate cholesterol administered intravenously in association with albumin, as a method to study reverse cholesterol transport (RCT) in humans by analyzing changes in the tracer activity in total plasma, lipoproteins and feces.

DETAILED DESCRIPTION:
The study will use 3H-cholesterol bound to albumin (particulate cholesterol) to assess the ability of HDL to transport cholesterol to the liver to be eliminated. This process is called Reverse Cholesterol transport and is one of the main mechanisms by which HDL protect against atherosclerotic cardiovascular disease. The availability of a method to assess RCT is important for the development of new drugs which affect RCT and may result in useful treatments for atherosclerosis.

This study will evaluate the use of radiolabeled particulate cholesterol administered intravenously in association with albumin, as a method to study reverse cholesterol transport (RCT) in humans by analyzing changes in the tracer activity in total plasma and lipoproteins. The study population is healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 70
2. Female subjects must be of non-childbearing potential. They must have been surgically sterilized at least 6 months prior to screening or be postmenopausal. Postmenopausal women must have no regular menstrual bleeding for at least 2 years prior to inclusion. .
3. Subjects must be in good overall health
4. Subjects must be able to comprehend and willing to provide a signed IRB approved Informed Consent Form.
5. Subjects must be willing to comply with all study-related procedures.

Exclusion Criteria:

1. Known cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease
2. History of diabetes mellitus or fasting glucose > 126 mg/dL at the screening visit
3. History of any other endocrine disease
4. History of a non-skin malignancy within the previous 5 years
5. Anemia; Hemoglobin less than 10 g/dL
6. Renal insufficiency as defined by creatinine ³ 1.3 mg/dl
7. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition
8. History of hypertension
9. Use of warfarin, or any known coagulopathy and /or elevated PT/PTT >1.5 x ULN
10. Self-reported history of HIV positive
11. Previous organ transplantation
12. Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests such as ALT or AST > 1x ULN, or self-reported history of positive Hepatitis B or Hepatitis C test result
13. Any major surgical procedure that occurred within the previous 3 months of the screening visit
14. Use of tobacco products currently or during the previous 30 days
15. History of drug abuse (< 3 years)
16. Regular use of alcoholic beverages (> 2 drinks/day)
17. Body mass index (BMI) > 30 kg/m2 or < 18.5 kg/m2
18. Participation in an investigational drug study within 6 weeks prior to the screening visit
19. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study will be excluded.
20. Use of lipid lowering drugs within the 6 weeks prior to dosing or during the study
21. Use of other prescription or non-prescription drugs (including vitamins and herbal supplements, but excluding replacement hormone therapy) within 2 weeks prior to dosing or during the study, however, acetaminophen up to 2g/day is acceptable.
22. Male subjects who plan to conceive a child within 3 months of the conclusion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in the tracer activity in total plasma and lipoproteins. | 10 minutes, Zero hour, 5, 10, 15, 30, 45 minutes, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 18, 24, 48, 72, 96 Hours

SECONDARY OUTCOMES:
Presence of the tracer in feces | Time zero to 96 Hour inclusive

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States